CLINICAL TRIAL: NCT00899158
Title: Role of Caspase-3, Phosphatidylinositol-3 Kinase (PI3K), and 3-methylhistidine (3-MH) in the Pathophysiology of Skeletal Muscle Loss in Weight-losing Pancreas Cancer Patients
Brief Title: Biological Markers in Patients With Pancreatic Cancer Experiencing Weight Loss
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE3204; P30CA043703 (NIH); CASE3204 (Other: Case Comprehensive Cancer Center); CWRU-020541
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Cachexia; Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; cachexia
MeSH Terms: conditions — Cachexia; Pancreatic Neoplasms | interventions — Immunologic Techniques; Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — During surgery, a muscle biopsy is performed and approximately 1 cm of rectus abdominous muscle is obtained for analysis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: immunologic technique
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Learning about biological markers in patients with pancreatic cancer and cachexia may help doctors predict patient outcome and may help the study of cancer in the future.

PURPOSE: This laboratory study is examining biological markers in patients with pancreatic cancer experiencing weight loss.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare levels of caspase-3 and phosphorylated Akt (pAkt) in the rectus abdominous muscle of patients with pancreatic cancer who are experiencing cachexia and are undergoing surgery for diagnosis or primary therapy with patients who have not lost weight and are undergoing abdominal surgery for nonmalignant conditions.
* Compare levels of urinary 3-methylhistidine (3-MH) in these patients.
* Evaluate possible correlations of caspase-3 activity, pAkt, and urinary 3-MH with early time to progression and subsequent lean body weight loss in patients with pancreatic cancer.
* Associate excretion of urinary 3-MH with higher levels of caspase-3 activity and pAkt to analyze the utility of 3-MH as a marker of skeletal muscle proteolysis.

OUTLINE: This is a pilot study.

During surgery, a muscle biopsy is performed and approximately 1 cm of rectus abdominous muscle is obtained for analysis. Caspase-3 activity and total/phosphorylated phosphatidylinositol-3 kinase and Akt are measured in muscle biopsies by western blot analysis. 3-methylhistidine activity is measured in urine samples.

After completion of study, patients with pancreatic cancer are followed postoperatively at 3 and 6 months.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis or suspicion of pancreatic cancer

    * Any stage disease allowed
    * At least 5% weight loss within the past 6 months
    * Scheduled to undergo exploratory surgery
  * Scheduled to undergo exploratory surgery for suspected nonmalignant condition

    * No weight loss OR weight loss due to specific reason (e.g., bowel obstruction, infection, or nausea/vomiting)
* No cancer diagnosis other than primary pancreatic carcinoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy ≥ 12 weeks
* No pacemakers or implanted defibrillators

PRIOR CONCURRENT THERAPY:

* Prior or concurrent chemotherapy and radiotherapy allowed
* Prior or concurrent biological therapy and surgery allowed
* At least 4 weeks since prior corticosteroids or anabolic steroids
* Other concurrent anticancer therapy allowed
* No concurrent corticosteroids or anabolic steroids, thalidomide, eicosapentaenoic acid (EPA), or Juven for weight loss

  * Concurrent steroids (i.e., antiemetics) associated with chemotherapy allowed
* No concurrent nutritional supplements with EPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle loss | Up to 6 months
Lean body mass | Up to 6 months
Time to progression | Up to 6 months
Caspase-3 levels | Up to 6 months
Phosphorylated Akt levels | Up to 6 months
Urinary 3-methylhistidine levels | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Brell, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States